CLINICAL TRIAL: NCT07147374
Title: Robotic Versus Open Surgery Following Neoadjuvant Therapy in Pancreatic Cancer: Evaluation of Safety and Oncologic Outcomes
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Robotic surgery
Record Dates: First submitted 2025-08-20; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Cancer; Neoadjuvant Therapy; Robotic Surgery
Keywords: Pancreatic cancer; Neoadjuvant therapy; Robotic surgery; Open surgery
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Robotic surgery: Patients who receive robotic pancreatic resection
- Open surgery: Patients who receive open pancreatic resection

SUMMARY:
The feasibility and safety of minimally invasive surgery in cases after neoadjuvant therapy were unclear. It is worth exploring the safety of robotic resection for pancreatic cancer following neoadjuvant therapy. The investigators investigated the comparative outcomes of robotic and open surgery in the management of pancreatic cancer after NAT, exploring the feasibility and safety of robotic procedures in complex cases of pancreatic cancer, and providing evidence-based guidance for clinical practice.

DETAILED DESCRIPTION:
Currently, most studies focus on upfront resectable pancreatic cancer, benign or low-grade malignant tumors, demonstrating that robotic surgery can shorten postoperative hospital stays, reduce intraoperative blood loss, and achieve oncological outcomes comparable to open surgery. The feasibility and safety of minimally invasive surgery in cases after NAT were unclear. Both the Miami international evidence-based consensus and the Brescia international validated European guidelines indicate that current data are insufficient to recommend minimally invasive approaches for pancreatic cancer resection following NAT, highlighting the need for additional research. Therefore, it is worth exploring the safety of robotic resection for pancreatic cancer following NAT.

The investigators investigated the comparative outcomes of robotic and open surgery in the management of pancreatic cancer after NAT, exploring the feasibility and safety of robotic procedures in complex cases of pancreatic cancer, and providing evidence-based guidance for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years.
* Received neoadjuvant chemotherapy.
* Postoperative pathology confirmed pancreatic cancer.
* Underwent either open or robotic surgery.

Exclusion Criteria:

* Intraoperative discovery of unresectable tumor or presence of distant metastasis.
* ASA score ≥ 4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pancreatic cancer who received neoadjuvant therapy and then received surgical resection
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Overall complication | Until the 90 days after surgery
  The complication occurred within 90 days after the surgery

SECONDARY OUTCOMES:
Clinically relevant postoperative pancreatic fistula | Until the 90 days after surgery
  Grade B or C pancreatic fistula within 90 days after surgery
Postoperative pancreatectomy hemorrhage | Until the 90 days after surgery
  Hemorrhage occurred within 90 days after surgery
Disease-free survival | Up to 2 years after the surgery
  The length of time from the completion of surgery until the recurrence of cancer, the occurrence of metastasis, death from any cause, or to the last follow-up.
Overall survival | Up to 2 years after surgery
  The length of time from the date of surgery to death from any cause or to the last follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Surgery, Peking Union Medical College Hospital (PUMCH), Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No